CLINICAL TRIAL: NCT03234010
Title: CSD170303: An Unblinded, Parallel, Randomized Study to Assess Nicotine Uptake in Smokers From Electronic Cigarettes
Brief Title: CSD170303: Study to Assess Nicotine Uptake in Smokers From Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD170303
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FT21092 Group (Experimental): 7 day at-home use of electronic cigarette FT21092 followed by a 2 day in-clinic period.
  Interventions: Other: FT21092
- FT21093 Group (Experimental): 7 day at-home use of electronic cigarette FT21093 followed by a 2 day in-clinic period.
  Interventions: Other: FT21093
- FT21096 Group (Experimental): 7 day at-home use of electronic cigarette FT21096 followed by a 2 day in-clinic period.
  Interventions: Other: FT21096
- FT21097 Group (Experimental): 7 day at-home use of electronic cigarette FT21097 followed by a 2 day in-clinic period.
  Interventions: Other: FT21097

INTERVENTIONS:
Other: FT21092 — An electronic cigarette
  Arms: FT21092 Group
Other: FT21093 — An electronic cigarette
  Arms: FT21093 Group
Other: FT21096 — An electronic cigarette
  Arms: FT21096 Group
Other: FT21097 — An electronic cigarette
  Arms: FT21097 Group

SUMMARY:
To determine the rate and amount of nicotine uptake with 10-minute ad libitum use of four different marketed electronic cigarettes. Furthermore, to measure overall product liking by subjects to assess potential willingness to seek out the Electronic Cigarette (EC) again in the future.

DETAILED DESCRIPTION:
This will be a single-center, randomized, open-label, parallel study during which up to 140 healthy adult subjects, consisting of 35 subjects per marketed EC product, will be enrolled. Subjects will be evaluated for plasma nicotine uptake, as well as overall product liking. The study will involve the use of four (4) marketed EC products in tobacco consumers who are exclusive smokers (i.e., naïve EC users) or dual users of cigarettes and ECs (i.e., intermittent EC users).

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an ICF and complete questionnaires written in English.
2. Generally healthy males and females, 21 to 60 years of age, inclusive, at Screening Visit.
3. Subjects must meet one (a or b) of the following tobacco use conditions:

   1. Exclusive cigarette smoker who self-reports smoking at least (≥) 10 cigarettes per day for at least 6 months prior to Screening Visit. Brief periods of abstinence more than 30 days prior to screening due to illness, quit attempt or clinical study participation will be allowed at the discretion of the Investigator.
   2. Dual user of combustible cigarettes and electronic cigarettes (EC) who self-reports:

   i. Smoking at least (≥) 10 cigarettes per day for at least 6 months prior to Screening Visit. Brief periods of abstinence more than 30 days prior to screening due to illness, quit attempt or clinical study participation will be allowed at the discretion of the Investigator and ii. Using a nicotine-containing cig-a-like EC or a tank system EC either daily or at least weekly for at least 3 months prior to Screening Visit.
4. Willing to be confined overnight and abstain from tobacco- and nicotine- containing product use for 12 hours prior to IP use through Study Discharge.
5. Willing to use assigned IP during the study according to protocol.
6. Expired breath carbon monoxide (ECO) level is ≥10 parts per million (ppm) at the Screening Visit and Study Day 1.
7. Positive urine cotinine test at the Screening Visit and Study Day 1.
8. No intent to quit smoking or vaping from the Screening Visit to Study Day 2.
9. Females must be willing to use a form of contraception acceptable to the Investigator from the time of signing informed consent until Study Discharge, or be surgically sterile for at least 90 days prior to the Screening Visit.

Exclusion Criteria:

1. Presence of clinically significant or unstable/uncontrolled acute or chronic medical conditions at the Screening Visit, as determined by the Investigator, that would preclude a subject from participating safely in the study (e.g., uncontrolled hypertension, diabetes, asthma or other lung disease, cardiac disease, neurological disease or psychiatric disorders) based on safety assessments such as clinical laboratory tests, pregnancy tests, medical history, and physical/oral examinations.
2. At risk for heart disease, as determined by the Investigator.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for 5 minutes.
4. Weight of ≤ 110 pounds.
5. Poor peripheral venous access.
6. Use of medicine for treatment of depression, unless on a stable dose for the past 6 months prior to screening and deemed clinically stable by the PI.
7. Current scheduled treatment for asthma within the past consecutive 12 months prior to screening. As needed treatment, such as inhalers, may be included at the PIs discretion pending approval from the medical monitor.
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and / or cryogenically removed.
9. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the Screening Visit.
10. History or presence of hemophilia or other bleeding disorders.
11. History or presence of clotting disorders with concomitant use of anticoagulants (e.g., clopidogrel [Plavix®], warfarin [Coumadin®, Jantoven®] or aspirin [> 325 mg/day]).
12. Participation in another clinical trial within (≤) 30 days prior to the time of consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of consent of the current study.
13. Positive test for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus antibody (anti-HCV).
14. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
15. Females ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
16. A positive urine drug screen without disclosure of prescribed corresponding concomitant medication(s) at the Screening Visit or on Study Day 1.
17. A positive alcohol breathalyzer result at the Screening Visit or on Study Day 1.
18. Employed by a tobacco or nicotine company, the study site, or handles tobacco or nicotine-containing products as part of their job.
19. Determined by the Investigator to be inappropriate for the study, including a subject who is unable to communicate or unwilling to cooperate with the clinical staff.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum baseline-adjusted nicotine plasma concentration) | -5, -0.5, 3, 5, 8, 10, 11, 12, 15, 20, 30, 60 Minutes
  To assess nicotine uptake with the start of a 10-minute ad libitum Investigational Product (IP) use period.
AUCnic0-60 | -5, -0.5, 3, 5, 8, 10, 11, 12, 15, 20, 30, 60 Minutes
  Area under the baseline-adjusted nicotine concentration-versus-time curve from time zero to 60 minutes after the start of a 10-minute ad libitum IP use period.

SECONDARY OUTCOMES:
Tmax | -5, -0.5, 3, 5, 8, 10, 12, 15 Minutes
  Maximum baseline-adjusted plasma nicotine concentration from time zero to 15 minutes after the start of IP use.
AUCnic0-15 | -5, -0.5, 3, 5, 8, 10, 12, 15 Minutes
  Area under the baseline-adjusted nicotine concentration-versus-time curve from time zero to 15 minutes after the start of IP use.
PLoverall | 13 Minutes
  Overall product liking (PL) is an additional measure of how much the subject likes the product, and is indicative of their potential willingness to seek out use of the product again at a later point in time; measured 13 minutes after the start of IP use.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Yoon, MSN, FNP-C, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No